CLINICAL TRIAL: NCT02989792
Title: A Study to Investigate the Genetic Variation of Dopamine Pathway Associated With the Observed Effects of a New Treatment in Former Studies in Patients With Chronic Pain
Brief Title: A Study to Investigate the Genetic Variation of Dopamine Pathway in Patients With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tools4Patient (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: T1001-03
Record Dates: First submitted 2016-12-05; First posted 2016-12-12 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Peripheral Neuropathy; Osteoarthritis
Keywords: pain
MeSH Terms: conditions — Peripheral Nervous System Diseases; Osteoarthritis; Pain | interventions — Blood Specimen Collection; Genotype

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unique study arm (Other)
  Interventions: Genetic: Blood sampling for genotyping; Other: Personality Questionnaires completion

INTERVENTIONS:
Genetic: Blood sampling for genotyping — Venous punction of maximum 10 millilitres
Other: Personality Questionnaires completion — Completion of the following questionnaires: Multidimensional Personality Questionnaire (MPSQ), Interpersonal Reactivity Index (IRI) and Behavioral inhibition system/ Behavioral activation systems (BISBAS) questionnaires

SUMMARY:
Patients having completed former trials T1001-01 or T1001-02 will undergo one blood sampling for genotyping purposes. In addition they will compete the personality questionnaires they had completed in the former trial.

ELIGIBILITY:
Inclusion Criteria:

* have completed T1001-01 or T1001-02 study (Visit 5 completed)
* are men or women of at least 18 years of age
* have given written informed consent approved by the relevant Ethics Committee governing the study sites

Exclusion Criteria:

* have any close relationship with the Investigators or the Sponsor
* are under legal protection, according to the national law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2017-10-05 (Actual); Study Completion 2017-10-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with Single Nucleotide Polymorphisms (SNPs) variation of catechol-O-methyltransferase | Time zero equals baseline
  SNPs will be analyzed with Sanger based genotyping or equivalent method
Number of participants with SNPs variation of monoamine oxidase | Time zero equals baseline
  SNPs will be analyzed with Sanger based genotyping or equivalent method
Number of participants with SNPs variation of dopamine B hydroxylase | Time zero equals baseline
  SNPs will be analyzed with Sanger based genotyping or equivalent method
Number of participants with SNPs variation of dopamine receptor 3 | Time zero equals baseline
  SNPs will be analyzed with Sanger based genotyping or equivalent method
Number of participants with SNPs variation of brain-derived neurotropic factor genes | Time zero equals baseline
  SNPs will be analyzed with Sanger based genotyping or equivalent method

SECONDARY OUTCOMES:
Number of participants with SNPs variation of tryptophan hydroxylase-2 | Time zero equals baseline
  SNPs will be analyzed with Sanger based genotyping or equivalent method
Number of participants with SNPs variation of 5-hydroxytryptamine transporter | Time zero equals baseline
  SNPs will be analyzed with Sanger based genotyping or equivalent method
Number of participants with SNPs variation of 5-hydroxytryptamine receptor 2A | Time zero equals baseline
  SNPs will be analyzed with Sanger based genotyping or equivalent method
Number of participants with SNPs variation of serotonin transporter gene-linked polymorphic region genes | Time zero equals baseline
  SNPs will be analyzed with Sanger based genotyping or equivalent method
Number of participants with SNPs variation of opioid receptor gene | Time zero equals baseline
  SNPs will be analyzed with Sanger based genotyping or equivalent method
Number of participants with SNPs variation of fatty acid amid hydrolase gene | Time zero equals baseline
  SNPs will be analyzed with Sanger based genotyping or equivalent method
Assessment of Cronbach alpha of the personality questionnaire used in this study and the former ones | Time zero equals baseline
  Cronbach's alpha between 0 and 1

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Pereira, Study Director — Tools4Patient
Locations (4):
- ATC SA, Liège, Belgium
- France (3):
  - CIC Clermont-Ferrand CHU G. Montpied, Clermont-Ferrand
  - Eurofins Optimed, Gières
  - Institut Curie, Paris